CLINICAL TRIAL: NCT02775825
Title: Quality of the End of Life Care for Adult Patients With Advanced Cancer in Saudi Arabia
Brief Title: Quality of the End of Life Care
Status: Completed | Type: Observational
Sponsor: National Guard Health Affairs (Other Government)
Responsible Party: Sponsor
Other Study IDs: C15/003/R
Record Dates: First submitted 2016-05-12; First posted 2016-05-18 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: survey

SUMMARY:
End-of life care is one of the principle components of cancer care. Measurement of the quality of care provided for end-of-life cancer patients is an important issue. Recently there has been an increased emphasis on measuring and monitoring the quality of cancer care for the purpose of improving clinical practice. Despite increasing attention paid to end-of-life care in recent years, many studies have described difficulties in the final phase of life, including problems with access to hospice, inadequate symptom management, care giving burdens, care mismatched with patient preferences, and inappropriate resource use. Measuring quality of life is an important issue for monitoring clinical practice and improving outcome. Although patient assessment is the best quality measure, it is impractical to measure the quality of end-of-life care because of the difficulties of accurate prognostication for end-of-life and many patients are too ill to provide assessments. In contrast, several recent studies developed quality indicators (QIs) of palliative and end-of-life care, which assess the quality from existing sources such as administrative data or medical chart data.

DETAILED DESCRIPTION:
Quality of care has been defined as the 'degree to which health services for individuals and populations increase the likelihood of desired health outcomes and are consistent with current professional knowledge'.The challenge remains, however, to define key indicators of quality of care, to link those indicators with health outcomes, and to establish reliable, valid, and timely measurements of the indicators.

The development of QIs is based on the assumption that there is available evidence or a consensus position that can be used to assess the quality of care provided. As many areas of health care interventions operate with a limited evidence base, it is often necessary to combine the existing evidence with consensus techniques; such techniques explore consensus among a group of experts to reach a final aggregate opinion, expert-based knowledge

A systematic review published in 2006 that reviewed literature and relevant websites from USA, Europe, Canada, and Australia concluded that there were limited tools to evaluate whether cancer patients receive effective supportive treatment. In response, the cancer-quality Assessing Symptoms Side Effects and Indicators of Supportive Treatment (ASSIST) measures were developed .These ninety two quality indicators (QIs) were developed for medical record abstraction using the RAND-UCLA QI development method; they cover assessment and treatment of pain and other symptoms as well as information and care planning. However there are a number of other indicators that can be studied these include intensive care unit (ICU) visit, Emergency (ER) visits and chemotherapy use close to death.

ELIGIBILITY:
Inclusion Criteria:

1. Documented confirmed cancer diagnosis.
2. 18 year or older.
3. Patients with advanced cancer (stage IV or with metastasis).
4. Any hospital admission within the last 30 days.

Exclusion Criteria:

1. Cancer patients admitted under care of other specialties other than oncology.
2. Patients who had a major surgery within one month of death, which required admission for more than 1 day under general anesthesia.
3. Patients who were following with other hospitals transferred and died within 3 days of admission.
4. Cancer diagnosis was made only on death certificate with no prior cancer diagnosis.
5. Patient died outside hospital.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with advanced cancer defined as patients who are 18 years or older with stage IV or metastatic disease at the last month of their life.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
To measure the quality of care provided by oncology department to adult patients with advanced cancer in the last month of their life using The Cancer Quality-ASSIST QI (Assessing Symptoms Side Effects and Indicators of Supportive Treatment | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdul Aziz Medical City for National Guard, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No